CLINICAL TRIAL: NCT04011332
Title: Nurse-led Integrated Care to Improve Quality of Life in COPD Patients With a Pulmonary Exacerbation
Brief Title: Nurse-led Integrated Care in COPD Patients With a Pulmonary Exacerbation
Acronym: NICCO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 2019-00797
Record Dates: First submitted 2019-07-04; First posted 2019-07-08 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: COPD Exacerbation
Keywords: integrated care; self-management

STUDY DESIGN:
Intervention Model Description: monocentric parallel cluster design with a baseline period
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental)
  Interventions: Other: Integrated Care Model
- Control Group (No Intervention)

INTERVENTIONS:
Other: Integrated Care Model — The patients who are hospitalised due to a COPD exacerbation will be aligned to a nurse-led integrated care model for three months. The model constitutes a bundle of interventions that are commonly known as key elements in COPD management. In addition, the ANP-Team (Advanced Nursing Practice-Team) will coordinate the different health professionals within the hospital and across transitions within the three months.
  Arms: Intervention Group

SUMMARY:
The aim of the study is to evaluate the effect and effectiveness of the nurse-led integrated care programme for the management of COPD (Chronic Obstructive Pulmonary Disease) exacerbations on patients' quality of life, rehospitalisation and exacerbation rate, illness-related emotional distress, selected health behaviours and cost-utility at three months. Furthermore, understanding barriers and facilitators to implementation success is of interest.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a confirmed diagnosis of COPD (GOLD 1-4)
* Hospitalisation due to a COPD exacerbation and decision to start with steroids and/or antibiotics (severe exacerbation)
* Age ≥ 18

Exclusion Criteria:

* Cognitive impairment (dementia, delirium)
* Not speaking German, French, Italian, English, Spanish, Portuguese, Serbian, Tamil, Hindi, Turkish or Slovakian

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2019-07-04 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Change in CRQ (Chronic Respiratory Questionnaire) scores | at week one and week 13
  Change in the four CRQ (Chronic Respiratory Questionnaire) subscores from week 1 to 13. The self-administered questionnaire version with standardised dyspnea questions (SAS) will be used. The questionnaire was developed for patients with chronic airflow limitations and comprises 20 items which assess four domains: 1) dyspnea, 2) fatigue, 3) emotional function and 4) mastery. The scoring scale ranges from 1 (extreme) to 7 (not at all) and will be assessed with a recall period of the past 2 weeks. A subscore for each domain (sum of items / number of items) will be calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schmid-Mohler G, Hubsch C, Braun J, Steurer-Stey C, Aregger C, Schaer DJ, Clarenbach C. Effect of a nurse-led integrated care intervention on quality of life and rehospitalisation in patients with severe exacerbation of COPD-a pilot study. Chron Respir Dis. 2024 Jan-Dec;21:14799731241291067. doi: 10.1177/14799731241291067. PMID 39407408